CLINICAL TRIAL: NCT00654238
Title: Phase II Study of BAY 43-9006 in Patients With Metastatic Thyroid Cancer
Brief Title: Phase II Trial of Sorafenib (Nexavar) in Patients With Advanced Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Marcia Brose, Associate Professor, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 802861; UPCC 03305; NCT00601783 (obsolete NCT alias)
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Differentiated Thyroid Cancer; Metastatic Poorly Differentiated Thyroid Cancer; Metastatic Anaplastic Thyroid Cancer; Metastatic Medullary Thyroid Cancer
Keywords: Thyroid Cancer; Anaplastic; Medullary; sorafenib
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Carcinoma, Medullary; Thyroid Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): This is a single arm study.
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — 400mg PO BID daily
  Other Names: Nexavar (Bayer)

SUMMARY:
The goal of this study is to determine the activity of sorafenib in patients with advanced (metastatic or recurrent) thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed thyroid cancer that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Patients may have received multiple treatments of radioactive iodine, one prior biologic treatment, and at least half of the patients will have had no prior chemotherapy for metastatic disease. At least 3 weeks must have elapsed since prior treatment.
* Measurable disease defined as at least one malignant lesion that can be accurately and serially measured in at least one dimension (longest diameter to be recorded), using a caliper (diameter > 10 mm) for superficial cutaneous disease, or using contrast-enhanced CT or spiral CT (diameter > 20 mm) for visceral or nodal/soft tissue disease.
* ECOG performance status < 2 (Appendix 1).
* Life expectancy greater than 3 months.
* Adequate organ function that has been determined within 7 days prior to enrollment, defined as:Leucocyte count > 3,000/uL; Absolute neutrophil count (ANC) > 1,500/mm3, platelets > 100,000/mm3, and hemoglobin > 9 g/dl; Serum creatinine < 1.5 times ULN, or 24-hour creatinine clearance > 75 cc/min. (Note: creatinine clearance need not be determined if the baseline serum creatinine is within normal limits); Serum bilirubin < 1.5 times ULN; serum glutamyloxaloacetic transaminase (SGOT) < 2.5 ULN; alkaline phosphatase < 2.5 times ULN; PT-INR/PTT < 1.5 x upper limit of normal.
* Intellectual, emotional, and physical ability to comply with oral medication.
* Ability to understand and the willingness to sign a written informed consent
* Patients with disease accessible for biopsy will be preferentially selected for participation in the study. Accessible disease includes lymph node metastases.
* Female patients of child-bearing potential must have a negative pregnancy test within 14 days before initiation of study drug dosing. Post-menopausal women must be amenorrheic for at least 12 months to be considered non-child-bearing potential. Male and female patients of reproductive potential must agree to use adequate contraception (i.e. hormonal or barrier method of birth control). throughout the study and for 3 months after the study.

Exclusion Criteria:

* Significant medical disease including: uncontrolled congestive heart failure; active symptoms of coronary artery disease, uncontrolled seizure disorder; active infection; uncontrolled diabetes mellitus; requirement for chronic corticosteroid treatment; requirement for concurrent immunosuppressive drug(s); active autoimmune disease.
* Organ allografts.
* Known HIV-infection (HIV testing is not required for participation).
* Pregnancy or lactation. Women of childbearing potential and sexually active males must be advised to take precautions to prevent pregnancy during treatment
* History of second cancer (except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for five or more years).
* Use of any experimental therapy within 3 weeks prior to baseline evaluations done prior to enrollment.
* Patients with carcinomatous meningitis are excluded from the study.
* Excluded therapies and medications, previous and concomitant:Anticancer chemotherapy or immunotherapy during the study or within 4 weeks prior to the first dose of the study drug; Radiotherapy for the treatment of a symptomatic (e.g. bone metastasis) as clinically indicated is allowed as long as it is not evidence of progressive disease (see 4.5.2); -Biological response modifiers, such as G-CSF, within 3 week prior to study entry. (G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator; however they may not be substituted for a required dose reduction); Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study; Investigational drug therapy outside of this trial during or within 4 weeks prior the screening assessment; Use of ketoconazole, itraconazole, and ritonavir; Use of carbamazepine, phenytoin, phenobarbital; Previous exposure to a Ras pathway inhibitor (including herceptin, EGFr inhibitors, farnesyl transferase inhibitors or MEK inhibitors); Use of grapefruit juice products; Use of cyclosporin;
* Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-02; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia S Brose, MD PhD, Principal Investigator — Unviersity of Pennsylvania - Abramson Comprehensive Cancer Center
Locations (1):
- University of Pennsylvania - Abramson Comprehensive Cancer Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib: This is a single arm study.
  sorafenib: 400mg PO BID daily
Period: Overall Study
Arm/Group | Sorafenib
Started | 59
Completed | 55
Not Completed | 4
Not completed — Screen Failures | 4

BASELINE CHARACTERISTICS:
Population: Four patients were deemed ineligible as a result of inadequate CBC and the establishment of an alternative diagnosis resulting from secondary pathology review.
Arm/Group | Sorafenib
Number analyzed (Participants) | 55
Age, Continuous [Median (Full Range); unit: years] | 63 [30 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 55
Histology subtype [Count of Participants; unit: Participants]
  DIfferentiated | 44
  Poorly Differentiated | 6
  Medullary | 3
  Anaplastic | 2
ECOG Performance Status at Baseline [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status is a well known classification system for patient performance status. The scale goes from 0 to 4. With 0 being fully active and functional and a 4 being 100% bedridden.
  Participants
    ECOG Performance Status 0 | 29
    ECOG Performance Status 1 | 26

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Efficacy (Best Response) of BAY 43-9006 (Objective Response Rate and Stable Disease) in Patients With Metastatic Thyroid Carcinoma.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Population: Responses were calculated by total enrolled to each group by histologic subtype.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib
Number analyzed (Participants) | 55
Participants
  Differentiated: number analyzed (Participants) | 44
  Differentiated: Complete Response | 0
  Differentiated: Partial response | 16
  Differentiated: Stable Disease | 22
  Differentiated: Progressive Disease | 1
  Differentiated: Not Evaluable for Response | 5
  Poorly Differenitated: number analyzed (Participants) | 6
  Poorly Differenitated: Complete Response | 0
  Poorly Differenitated: Partial response | 2
  Poorly Differenitated: Stable Disease | 1
  Poorly Differenitated: Progressive Disease | 1
  Poorly Differenitated: Not Evaluable for Response | 2
  Medullary: number analyzed (Participants) | 3
  Medullary: Complete Response | 0
  Medullary: Partial response | 1
  Medullary: Stable Disease | 2
  Medullary: Progressive Disease | 0
  Medullary: Not Evaluable for Response | 0
  Anaplastic: number analyzed (Participants) | 2
  Anaplastic: Complete Response | 0
  Anaplastic: Partial response | 0
  Anaplastic: Stable Disease | 0
  Anaplastic: Progressive Disease | 1
  Anaplastic: Not Evaluable for Response | 1

2. Secondary Outcome: Median Progression Free Survival in Patients Receiving BAY 43-9006 (Sorafenib).
Description: This is the result of the Kaplan Meier analysis of all patients treated with sorafenib
Time Frame: as for outcome 1
Population: Of the 59 patients that were consented, four patients were deemed ineligible as a result of inadequate CBC and the establishment of an alternative diagnosis resulting from secondary pathology review. Therefore the total number of patients analyzed going forward was 55.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Progression Free Survival For Entire Study (55 Total Patients): This is based on Kaplan Meier estimate
Arm/Group | Progression Free Survival For Entire Study (55 Total Patients)
Number analyzed (Participants) | 55
weeks | 77 [60 to 96]

ADVERSE EVENTS:
Time Frame: 5 Years
Arm/Group | Sorafenib
All-Cause Mortality (participants affected / at risk) | 36/55
Serious Adverse Events (participants affected / at risk) | 4/55
Other Adverse Events (participants affected / at risk) | 43/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (N=55)
Deep Vein Thhrombosis (Blood and lymphatic system disorders) | 2 (2) — Two patients had DVT Grade 3
Cerebral Vascular Accident/Stroke (Nervous system disorders) | 2 (2) — Cerebral Vascular Accident and or Stroke
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (N=55)
Hand Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 43 (43) — All Grades
Rash (Skin and subcutaneous tissue disorders) | 41 (41) — All Grades
Diarrhea (Gastrointestinal disorders) | 29 (29) — All Grades
Alopecia (Skin and subcutaneous tissue disorders) | 25 (25) — All Grades
Stomatitis/Mucositis (Gastrointestinal disorders) | 18 (18) — All Grades
Fatigue (General disorders) | 15 (15) — All Grades
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11) — All Grades
GI Discomfort (Gastrointestinal disorders) | 9 (9) — All Grades
Hypertension (Vascular disorders) | 8 (8) — All Grades
Squamous Cell Carcinoma of the Skin (Skin and subcutaneous tissue disorders) | 8 (8) — All Grades
Anorexia and Weight Loss (Metabolism and nutrition disorders) | 7 (7) — All Grades
Hepatic Lab Abnormalities (Gastrointestinal disorders) | 1 (1) — All Grades

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No